CLINICAL TRIAL: NCT04477577
Title: First Heroes: Engaging Fathers in the First 1000 Days
Acronym: First Heroes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elsie Taveras, MD, Division Chief, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019P003739
Record Dates: First submitted 2020-07-08; First posted 2020-07-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2024-04

CONDITIONS: Obesity, Childhood; Overweight and Obesity; Social Determinants of Health; Physical Activity; Feeding Behavior; Sleep; Diet Habit
Keywords: Overweight; Obesity; Social Determinants of Health; Maternal-Child Health
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity; Motor Activity; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New Parent Intervention (Experimental)
  Interventions: Behavioral: New Parent Intervention
- Safety Control (Active Comparator)
  Interventions: Behavioral: Safety Control

INTERVENTIONS:
Behavioral: New Parent Intervention — This arm will receive the Obstetric and Pediatric primary care provided within MGH obstetric and pediatric primary care practices, with additional active and targeted engagement of new parents by a health coach.
  Arms: New Parent Intervention
Behavioral: Safety Control — This arm will receive the Obstetric and Pediatric primary care provided within MGH obstetric and pediatric primary care practices, with additional infant safety education materials.
  Arms: Safety Control

SUMMARY:
The First Heroes study plans to influence weight and health trajectories, modify disease risk, and improve health care services for mother-father-infant triads from racial/ethnic minority and health disparity populations.

This study is a two-arm, randomized controlled trial recruiting from Massachusetts General Hospital (MGH) obstetrics practices. This study will enroll 250 father-mother dyads in the second trimester of pregnancy and intervene through their offspring's 1-year birthday. Each mother-father dyad participating will be randomly assigned to one of two arms: 1. Obstetric and Pediatric Standard of Care + New Parent Engagement Intervention Arm or; 2. Obstetric and Pediatric Standard of Care + Safety Control Arm.

ELIGIBILITY:
Inclusion Criteria:

* Parental dyads must meet the following criteria:
* Pregnant females and father of the baby, both aged ≥ 18 years
* Singleton pregnancy
* Planned involvement during the first year of the child's life
* Planning to receive post-partum and pediatric care for child at any pediatric practice within the MassGeneral Brigham (Partners) Healthcare system
* Ability to speak in English or Spanish
* Capable of giving consent

Exclusion Criteria:

* Dyads whose unborn child is found to have a severe defect or comorbidity upon 18-20 week ultrasound.
* Mothers who intend on raising a child alone without any participation from the father of the child.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of rapid infant weight gain | Birth to child age 6 months
  Weight-for-length z-score
Prevalence of rapid infant weight gain | Birth to child age 12 months
  Weight-for-length z-score
Prevalence of overweight in infants | Birth to child age 12 months
  Weight-for-length ≥97.7th percentile based on World Health Organization standards
Prevalence of overweight in infants | Birth to child age 12 months
  Weight-for-length ≥95 percentile based on Center for Disease Control

SECONDARY OUTCOMES:
Maternal post-partum weight retention | Child birth to 6-month postpartum
  Weight in kilograms
Maternal post-partum weight retention | Child birth to 12-month postpartum
  Weight in kilograms
Maternal diet | Baseline to 6-month postpartum
  Average weekly intake of fruits and vegetables
Maternal diet | Baseline to 12-month postpartum
  Average weekly intake of fruits and vegetables
Maternal physical activity | Baseline to 6-month postpartum
  Days per week physically active for at least 30 minutes per day
Maternal physical activity | Baseline to 12-month postpartum
  Days per week physically active for at least 30 minutes per day
Maternal adherence to preventive health services | Baseline to 12 months post-partum
  Number of preventative care visits attended
Paternal Mean Body Mass Index | Baseline to 6-month postpartum
  Mean change in paternal BMI calculated by weight in kilograms and height in meters to report BMI in kg/m^2.
Paternal Mean Body Mass Index | Baseline to 12-month postpartum
  Mean change in paternal obesity calculated by weight in kilograms and height in meters to report BMI in kg/m^2.
Paternal prevalence of obesity | Baseline to 12-month postpartum
  Prevalence of BMI≥30 kg/m2 calculated by weight in kilograms and height in meters.
Paternal adherence to preventive health services | Baseline to 12-month post-partum
  Number of preventative care visits attended
Paternal diet | Baseline to 6 months post-partum
  Average weekly intake of fruits and vegetables
Paternal diet | Baseline to 12 months post-partum
  Average weekly intake of fruits and vegetables
Paternal physical activity | Baseline to 6 months post-partum
  Days per week physically active for at least 30 minutes per day
Paternal physical activity | Baseline to 12 months post-partum
  Days per week physically active for at least 30 minutes per day
Parental perceived stress | 6 month post-partum
  Perceived Stress Scale - 4-item validated scale
Prevalence of parental post-partum depression | 6 month post-partum
  Patient Health Questionnaire 2 (PHQ-2)
Prevalence of parental post-partum depression | 12 month post-partum
  Patient Health Questionnaire 2 (PHQ-2)
Prevalence of breastfeeding initiation | 6 months post-partum
  Self-reported response questionnaire
Infant introduction of solid foods | 6 months post-partum
  Self-reported response questionnaire

OTHER OUTCOMES:
Family enrollment in food assistance programs during intervention period | Baseline to 12 months post partum
  Yes/No response options for program enrollment in WIC/SNAP
Family housing insecurity during intervention period | Baseline to 12 months post partum
  National Survey of American Families - 2-item validated scale
Family food insecurity during intervention period | Baseline to 12 months post partum
  Hager 2-question validated scale

CONTACTS AND LOCATIONS:
Overall Officials: Elsie Taveras, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silver SR, Whooten RC, Kwete GM, Farrar-Muir H, Cournoyer RN, Barth EA, Kotelchuck M, Taveras EM. Stakeholder engagement in developing a father-inclusive early life obesity prevention intervention: First Heroes. BMC Pregnancy Childbirth. 2022 May 27;22(1):443. doi: 10.1186/s12884-022-04759-z. PMID 35624421
- [Background] Whooten RC, Kwete GM, Farrar-Muir H, Cournoyer RN, Barth EA, Kotelchuck M, Taveras EM. Engaging fathers in the first 1000 days to improve perinatal outcomes and prevent obesity: Rationale and design of the First Heroes randomized trial. Contemp Clin Trials. 2021 Feb;101:106253. doi: 10.1016/j.cct.2020.106253. Epub 2020 Dec 17. PMID 33340750
- [Background] Whooten RC, Kotelchuck M, Gonzalez AVC, Johnson N, Kwete G, Luo M, Muir HF, Barth EA, Smith N, Taveras EM. Expectant fathers' health behaviors, infant care intentions, and social-emotional wellbeing in the perinatal period: A latent class analysis and comparison to mothers. Prev Med Rep. 2023 Aug 26;36:102375. doi: 10.1016/j.pmedr.2023.102375. eCollection 2023 Dec. PMID 37719794